CLINICAL TRIAL: NCT01753206
Title: Observational Study to Investigate Resistant Hypertension Prevalence Among the Hypertensive Patients Who Have Been Treated in Korean General Hospitals
Brief Title: Observational Study to Investigate Resistant Hypertension Prevalence in Korean General Hospitals
Acronym: Teveten_RH
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD_EPR_OS2012
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Objectives The study is to identify prevalence, demography and clinical characteristics of patients with resistant hypertension among hypertensive patients who have been treated in general hospitals in Korea from Jan 2012 to Jun 2012.

* Diagnosis of resistant hypertension: In case of clinic blood pressure exceeding the boundary of systolic blood pressure at 140mmHg and diastolic blood pressure at 90mmHg (hereinafter refer to as 140/90mmHg) (130/80mmHg for patients with diabetes mellitus or chronic renal disease) despite triple antihypertensive therapy at optimal dose may be diagnosed as resistant hypertension. Antihypertensive medications used include diuretics. Resistant hypertension may also be diagnosed when clinic blood pressure has reached the target value but quadruple or more of antihypertensives are used.
* Diagnosis of controlled hypertension: Patients whose clinic blood pressure equals to 140/90mmHg (130/80mmHg for patients with diabetes mellitus or chronic renal disease) or less with the administration of antihypertensives at optimal dose may be diagnosed as controlled hypertension.

DETAILED DESCRIPTION:
Primary Objective:

Prevalence in patients with resistant hypertension among hypertensive patients who have been treated in Korean general hospitals

Secondary Objectives:

Analysis of correlation in patients with resistant hypertension and patients with controlled hypertension who received triple antihypertensive therapy in terms of demography, clinical characteristics and other factors

1. Demographic data (age, sex, and body mass index)
2. Clinical characteristics

   * Vital signs
   * Lifestyles (history of drinking, smoking, and exercise)
   * Family history (hypertension, diabetes mellitus, dyslipidemia, cardiovascular disease, renal/adrenal disease, cerebrovascular disease, and respiratory disease)
   * Concurrent diseases (diabetes mellitus, dyslipidemia, cardiovascular disease, renal/adrenal disease, cerebrovascular disease, respiratory disease, and others)
   * History of antihypertensive therapy (past and present)
   * Medication compliance of antihypertensives
   * Concomitant medications

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed of hypertension and in 20 years of age or older at the time of participating the study
2. Patients visiting the medical institution during the period of 01 2012 ~ 06 2012 and who have received triple or more of antihypertensive therapy including diuretics (all different classes one another) at the time of the investigation.
3. Patients who signed the informed consent form for data use before undergoing the study procedures.
4. Patients who have capability and are willing to understand and fill in the questionnaire used in this study or who have a representative to fill in the questionnaire in case of lacking the capability.

Exclusion Criteria:

1. Patients who fail to meet the inclusion criteria.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1579 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of resistant hypertension | up to 6 months
  Prevalence of resistant hypertension will be estimated, and its 95% confidence interval will be calculated. In addition, proportion of controlled hypertensive patients and its 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Analysis of correlation in patients with resistant hypertension and patients with controlled hypertension who received triple antihypertensive therapy in terms of demography, clinical characteristics and other factors | up to 6 months
  Clinical characteristics in subjects diagnosed of resistant hypertension and those diagnosed of controlled hypertension will be described in summary.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu, South Korea